CLINICAL TRIAL: NCT06127225
Title: The Effect of Proliverenol Supplementation on Liver Function in Patients With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Proliverenol Supplementation for Non-Alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: PT Equilab International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR.079/EQL/2021
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD; Proliverenol
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment 1 (Experimental): 1 caplet of Proliverenol 500 mg twice daily
  Interventions: Drug: Proliverenol
- Treatment 2 (Experimental): 2 caplets of Proliverenol 500 mg once daily
  Interventions: Drug: Proliverenol
- Treatment 3 (Experimental): 2 caplets of Proliverenol 500 mg twice daily
  Interventions: Drug: Proliverenol
- Treatment 4 (Placebo Comparator): 2 caplets of Placebo daily
  Interventions: Drug: Placebo caplets of Proliverenol

INTERVENTIONS:
Drug: Proliverenol — 1 caplet of Proliverenol 500 mg twice daily 2 caplets of Proliverenol 500 mg once daily 2 caplets of Proliverenol 500 mg twice daily
  Arms: Treatment 1; Treatment 2; Treatment 3
Drug: Placebo caplets of Proliverenol — 2 caplets of Proliverenol Placebo daily
  Arms: Treatment 4

SUMMARY:
This is a 4-arm, prospective, randomized, double-blind, double-dummy, and placebo-controlled clinical study comparing Proliverenol at a dose of 500 mg twice daily; Proliverenol at a dose of 1000 mg once daily; Proliverenol at a dose of 1000 mg twice daily; and Placebo two caplets daily for a 12-week course of therapy.

Proliverenol is a bioactive fraction derived from the dried fruit of Phaleria macrocarpa (Scheff.) Boerl (Thymelaeaceae). Proliverenol possesses a hepatoprotective activity via anti-inflammation, DNA repairing, and the antiapoptosis properties.

DETAILED DESCRIPTION:
There will be 4 groups of treatment; each group will consist of 20 subjects with the treatment regimens for 12 weeks:

Treatment I : 1 caplet of Proliverenol 500 mg twice daily Treatment II : 2 caplets of Proliverenol 500 mg once daily Treatment III : 2 caplets of Proliverenol 500 mg twice daily Treatment IV : 2 caplets of Placebo daily

Study subjects will be asked to come to the clinic every 4-week interval throughout the study period.

Subjects will be evaluated for treatment efficacy at baseline and at interval of 4 weeks over the 12-week course of therapy. Throughout the 12-week therapy, subjects should record the product consumption and adverse event occurred during the study in the provided Patient's Diary.

The safety profile of study medication other than vital signs and adverse event will be measured at baseline and end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Male or female subjects with age of 18 years or older at screening.
3. Diagnosed as NAFLD with liver ultrasonography (USG). Patients with bright liver appearance based on USG, will be followed by CAP examination. Steatosis is defined if CAP >263 dB/m
4. Presence of hepatic impairment, defined as any of serum ALT level > ULN
5. Able to take oral medication.

Exclusion Criteria:

1. Suspected positive COVID-19 based on clinical symptoms or SARS-COV-2 antigen test
2. Pregnancy and lactation period.
3. Suspected alcoholic liver disease
4. History of or presence of autoimmune liver diseases
5. Presence of Bilirubin level > 2x ULN
6. Uncontrolled Diabetes Mellitus with HbA1c ≥ 9.0%
7. History or presence of significant/advanced CV, metabolic, acute or chronic infectious diseases, including viral hepatitis (B and C), or malignancy.
8. Suspected cirrhosis as supported by biochemical profile (PLT count, albumin)
9. Presence of severe renal dysfunction
10. Current or regular use of drug-induced hepatotoxicity, such as: such as non-steroidal anti-inflammatory drugs (NSAIDs), antibiotics, anti-epileptic drugs (e.g. carbamazepines, phenytoin, barbiturates), or anti-tuberculous drugs other than the investigational product
11. Current or regular use of herbal medicines with hepato-protective properties
12. Known or suspected hypersensitivity to the trial product or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Changes of serum ALT levels | 4, 8, and 12 weeks
  Changes of serum ALT levels from baseline to Week 4, 8, and 12 of study treatment
Changes of serum AST levels | 4, 8, and 12 weeks
  Changes of serum AST levels from baseline to Week 4, 8, and 12 of study treatment

SECONDARY OUTCOMES:
USG examination for Controlled Attenuated Parameter (CAP) | 0 and 12 weeks
  USG examination for Controlled Attenuated Parameter (CAP) measurement will be performed on baseline and week 12 of study treatment
USG examination for Transient elastography (TE) | 0 and 12 weeks
  USG examination for Transient elastography (TE) measurement will be performed on baseline and week 12 of study treatment
Ratio of Aspartate transaminase (AST) to alanine transaminase (ALT) serum levels | 4, 8, and 12 weeks
  Ratio of Aspartate transaminase (AST) to alanine transaminase (ALT) serum levels at Week 4, 8, and 12 of study treatment
Liver function (GGT and AP) | 0 and 12 weeks
  Concentration of serum gamma-glutamyl transpeptidase (GGT) and alkaline phosphatase (AP) at Baseline and at the End of study
Liver function (Bilirubin) | 0 and 12 weeks
  Concentration of total bilirubin at Baseline and at the End of study
Lipid profile (Total cholesterol, LDL, HDL, triglyceride) | 0 and 12 weeks
  Concentration of total cholesterol, LDL, HDL, triglyceride at Baseline and at the End of study
Renal function (Ureum and creatinine) | 0 and 12 weeks
  Level of ureum and creatinine at Baseline and at the End of study
Hematology test | 0 and 12 weeks
  Hematology test (especially leucocyte and platelet counts) at Baseline and at the End of study
Adverse events | 4, 8, and 12 weeks
  Adverse event, will be observed throughout the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Irsan D. Hasan, MD, SpPD, KGEH, Principal Investigator — Division of Hepatology, Departement of Internal Medicine Faculty of Medicine, University of Indonesia Dr. Cipto Mangunkusumo Hospital
Locations (1):
- Division of Hepatology, Dr. Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia